CLINICAL TRIAL: NCT03324620
Title: Cost-effectiveness of a Functional and Respiratory Rehabilitation Intervention in Patients Who Receive an Allogeneic Hematopoietic Stem Cell Transplantation (HSCT).
Brief Title: Effectiveness Rehabilitation Hematopoietic Transplantation (ovERsHOT)
Acronym: ovERsHOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Yolanda Torralba Garcia, Clinical investigator. BSN., Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2012-7705
Record Dates: First submitted 2017-09-19; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: physiotherapy; nurse; Cost effectiveness; Activities of Daily Living; exercise tolerance; Allogeneic; Quality of Life; Rehabilitation; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Mixed study. Retrospective control group.
Masking Description: 86 patients in experimental group. 104 patients retrospectively collected from the inclusion of the first patient of the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre active HSCT (Experimental): Candidates for transplantation of hematopoietic progenitors since May 12, 2012, regardless of sex and age, who agree to participate in the study and sign informed consent.
  In the pre-transplantation visit with the physiotherapist: Measures of muscle mass and strength, quality of life questionnaires, program presentation, fitness assessment and lifestyle determination. The exercises will be personalized, stimulating your practice before admission and involving the family. During admission, the team will encourage the patient to remain active by adapting to the symptoms. At discharge, measures of resistance, exercise tolerance and quality of life at discharge, in the month after discharge, 3 months after discharge, 6 months after discharge and 12 months after discharge.
  Interventions: Other: Specific program functional and respiratory rehabilitation
- control group (No Intervention): Patients' candidates for transplantation of hematopoietic progenitors prior to May 12, 2012, regardless of gender and age, who meet the inclusion criteria and are collected correlatively until completing 104 subjects.
  Clinical history review to calculate the days of hospitalization in the different hospitalization units during the transplant. As well as the number and type of complications and the use of health resources. Status vitae. Baseline review of functional tests and exercise tolerance.

INTERVENTIONS:
Other: Specific program functional and respiratory rehabilitation — It is a question of introducing a small program of physical activation pre-transplantation of hematopoietic progenitors, to continue developing it during the hospitalization and to use the functional measurements as a measure of its impact, as well as the different quality of life questionnaires.
  Arms: pre active HSCT

SUMMARY:
The objective of the study is to evaluate the benefits and costs of a comprehensive rehabilitation program (physical, psychological, social and educational) for patients receiving hematopoietic stem cell transplantation (HSCT). It is a prospective longitudinal study with a control group. Patients will be included who will perform a transplant in the hospital environment. The variables of the study will be: number and type of complications, days of hospitalization, readmissions, economic cost of the program, exercise tolerance, assessment of muscular atrophy, health related quality of life, knowledge and self-management of the disease, all of them adjusted for the variables age, sex and hematological disease, as well as comorbidities. The evaluations will be performed before transplantation (between one and three months before), during the conditioning phase (intensive chemotherapy), before discharge, after immediate discharge and after discharge up to one year. The nursing team will perform the patient's therapeutic education, stimulation for physical activity, as well as evaluation and follow-up measures. Early detection of the needs of the rest of the rehabilitation team will be carried out. There will be a support function for the physiotherapist in regard to physical activity. In Spain there is no interdisciplinary team that provides comprehensive care and rehabilitation to this type of patients and few studies are dedicated to rehabilitation beyond physiotherapy as a preventive tool for future disabilities.

DETAILED DESCRIPTION:
Working hypothesis

* 1. Patients who receive a Hematopoietic Stem Cell Transplantation (HSCT) who follow a comprehensive rehabilitation program, have fewer post-transplant complications, reduce the number of hospital stay days, and return to their daily lives more quickly.
* 2. The economic costs derived from the incorporation of the rehabilitation program will be lower than the savings caused by the decrease in complications, hospital stay and consumption of health resources.

Goals

Main objectives

* To evaluate the quality of life related to health in the hematological patient who has received a HSCT and on which a new preventive functional rehabilitation intervention (other than physiotherapy) is applied.
* To compare the number and type of respiratory and other complications after HSCT among the intervention group compared to a control group.
* Estimate the effects of the rehabilitation program on tolerance to exercise in the short, medium and long term, as well as detect the change in lifestyle if this occurred.

Secondary objectives

* Evaluate and compare the days of hospital stay and the time elapsed in each of the specialized units (insulation, Intensive Care Unit, single room with High Efficiency Particulate Air, (HEPA filter).
* To qualify the economic costs of the physiotherapy intervention within the rehabilitation program, the complications and the days of hospitalization.
* To evaluate the incidence of muscular atrophy and the level of tolerance to the effort as indicative of physical deconditioning and sedentary lifestyle.
* Measure the amount of symptoms, or the frequency of them: pain (measured by visual analog scale for pain (VAS), nausea / vomiting, insomnia, anxiety, anorexia ...)

Methodology

This is a prospective experimental study with a control group prior to the start of the intervention, which will include 190 participants. The sample size was calculated using a 95% confidence level and considering a positive and negative variability of 50% since there are no previous studies applying this methodology and taking into account the high mortality associated with the infection that oscillates between 35 and 50% according to the studies. The subjects will be treated in the hospital setting in airtight rooms with HEPA filters. Patients will be collected correlatively from the moment they enter the transplant program and sign informed consent. The control group will be collected retrospectively, from the day 1 of the startup of the program to 75, after verifying that they do not meet any inclusion criteria. Recruitment and incorporation into the study will be continuous according to the appearance of cases that meet the inclusion criteria.

The study will include patients receiving HSCT for the next 2 years from the study start date and will be followed and evaluated for a period of one year after transplantation.

Outcomes:

Quality of life, post-transplant complications, especially respiratory, capacity for exercise tolerance, muscular atrophy, onset of sleep disorders, days of stay in different hospital units, cost of interventions: physiotherapy, treatment of complications, and program rehabilitation. Mortality related to the transplantation, which covers any lethal complication from the moment of conditioning and without intervening the patient's underlying disease, that is, the progression of the same. Assess adherence to the program and evaluation and knowledge acquired by the patient.

Measurements:

To make the measurements, use:

* Bioimpedance analysis body composition (BIA), (Quantum X, RJL-Systems instruments™, Mi, USA): This test is performed on the patients in the intervention group at baseline, at discharge from hospital for transplantation, at the month of discharge, and at 3, 6, and 12 months, in order to assess their body composition, their fat mass and their muscle mass.
* Six-minute-walk test (to complement the assessment of exercise tolerance): This test is performed on the patients in the intervention group at baseline, at discharge from hospital for transplantation, at the month of discharge, and at 3, 6, and 12 months, in order to assess the exercise tolerance described in meters traveled, percentage of normality, symptomatology (dyspnea / fatigue of legs), and heart rate recovery. The abrupt weight changes in this population will be decisive for the interpretation of these data.
* Muscle strength test (handgrip (Jamar™ Dynamometer, Preston, Jackson, Mi, USA) and 1RM): This test is performed on the patients in the intervention group at baseline, at discharge from hospital for transplantation, at the month of discharge, and at 3, 6, and 12 months, in order to assess the strength in upper limbs at different times of process.
* Functional Assessment of Cancer Therapy questionnaires (FACT) validated in Spanish, to measure quality of life associated with the disease (lymphoma (LYM), leukemia (LEU), multiple myeloma (MM), Bone marrow transplantation (BMT); fatigue, anorexia): This test is performed on the patients in the intervention group at baseline, at discharge from hospital for transplantation, at the month of discharge, and at 3, 6, and 12 months in order to evaluate subjectively different aspects of health: functional, physical, emotional, as well as other concerns and symptoms associated with the process.
* Physical activity questionnaire for adult subjects -Modified Baecke Questionnaire™- (to measure the sedentary lifestyle): This test is performed on the patients in the intervention group at baseline, at discharge from the transplant hospital, at the month of discharge, and at 3, 6, and 12 months, in order to subjectively assess physical activity which subjects can develop during the first year of the transplant, and if there are limitations due to complications or readmissions.
* Anxiety-depression assessment (HAD) questionnaire. This test is performed on patients in the intervention group at baseline, at discharge from the transplant hospital, at the month of discharge, and at 3, 6, and 12 months, in order to assess the role of anxiety and depression at different times of the transplant and its follow-up in one year.
* Pittsburgh Sleep Quality Index. This test is performed on the patients in the intervention group at baseline, at discharge from the transplant hospital, at the month of discharge, and at 3, 6, and 12 months, in order to assess the subjective quality of sleep in these patients during the transplant period and their follow-up for one year. It is intended to evaluate the previous present difficulties, the use of hypnotics or other drugs used, and the need for continuity of treatments, as well as the effectiveness of them. The quality of sleep in hospitalized patients is highly documented, but it is not present in this type of patients nor is there any longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant hemopathies candidates for HSCT.
* controlled pain.
* who sign informed consent.

Exclusion Criteria:

* Severe musculoskeletal or neurological alterations prior to HSCT.
* Severe psychiatric problems.
* Language barrier.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2012-05-12 (Actual); Primary Completion 2012-05-12 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Cost of interventions assesed by the cost of hospitalization for HSCT | Admission
  For the calculation the days of hospitalization in each hospitalization unit care are counted. Then, the total number of days spent in each unit (D): (intensive care unit, ICU (A), isolation chamber (B), single room (C).
  The cost of hospitalization for HSCT: (a: price / day in the ICU, b: price / day in isolation chamber, c: price / day in single room, in euros). Dd = (Aa) + (Bb) + (Cc), in euros.
Cost of interventions assesed by the cost incorporation of a physiotherapist into the team | Admission
  To calculate the cost, a physiotherapist will be hired 4 hours / day for the intervention group. Day of hospitalization for the transplant (D) multiplied by the cost per day of the physiotherapist (euros).
Cost of interventions assesed by the number (number), characteristics and incidence of the immediate complications of HSCT | Admisssion
  Incidence expressed as a percentage. Comparison between the two groups (total number and percentage)
Cost of interventions assesed by antimicrobials used in infectious complications and chemotherapy conditioning. | Admission
  expressed in euros

SECONDARY OUTCOMES:
Adherence to the program and evaluation of the knowledge acquired by the patient. | Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  At each visit the patient will be purposely questioned about adherence to the exercise program. Non-adherence data will be collected, such as "I am bored with exercises", "I am very tired or have a lot of symptoms", "I am depressed or sad". In addition, each interview will gather training / information data explained in the previous interview. For example: Visit 1: adherence to treatment. Immunosuppressants. Importance of water intake. Neutropenic diet.
Referred quality of life: quality of life as assessed by the FACT (Functional Assessment of Cancer Therapy) leukemia questionnaire (Scale info can be included in the description.) | Admission.
  Initially, the FACT (Functional evaluation of cancer therapy) questionnaire will be used according to the baseline disease: FACT_leukemia; (range 0-176 units on a scale). The highest scores in each category translate into a better quality of life. The questionnaire is divided into 4 sections: physical status (range 0-28 units), family and social environment (range 0-28 units), emotional state (range 0-24 units), operating capacity (range 0-28) and other concerns - leukemia-specific (range 0-68). The total score FACT_leukemia is the sum of all the sections. Also in the subsections the higher the score the better the perceived quality of life. The physical, environmental, emotional and functional capacity is common in all FACT questionnaires used, which allows comparing this aspect between subjects.
Referred quality of life: quality of life as assessed by the FACT (Functional Assessment of Cancer Therapy) lymfhoma questionnaire (Scale info can be included in the description.) | Admission.
  Initially, the FACT (Functional evaluation of cancer therapy) questionnaire will be used according to the baseline disease: FACT_lymphoma; (range 0-168 units on a scale). The highest scores in each category translate into a better quality of life.
  The questionnaire is divided into 4 sections: physical status (range 0-28 units), family and social environment (range 0-28 units), emotional state (range 0-24 units), operating capacity (range 0-28) and other concerns - lymfoma-specific (range 0-60). The total score FACT_lymfoma is the sum of all the sections. Also in the subsections the higher the score the better the perceived quality of life. The physical, environmental, emotional and functional capacity is common in all FACT questionnaires used, which allows comparing this aspect between subjects.
Referred quality of life: quality of life as assessed by the FACT (Functional Assessment of Cancer Therapy) multiple myeloma questionnaire (Scale info can be included in the description.) | Admission.
  Initially, the FACT (Functional evaluation of cancer therapy) questionnaire will be used according to the baseline disease: FACT_multiple myeloma; (range 0-164 units on a scale). The highest scores in each category translate into a better quality of life.
  The questionnaire is divided into 4 sections: physical status (range 0-28 units), family and social environment (range 0-28 units), emotional state (range 0-24 units), operating capacity (range 0-28) and other concerns - myeloma-specific (range 0-56). The total score FACT_multiple myeloma is the sum of all the sections. Also in the subsections the higher the score the better the perceived quality of life. The physical, environmental, emotional and functional capacity is common in all FACT questionnaires used, which allows comparing this aspect between subjects.
Referred quality of life: quality of life as assessed by the FACT (Functional Assessment of Cancer Therapy) Bone marrow transplant (Scale info can be included in the description.) | Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  The questionnaire is divided into 4 sections: physical status (range 0-28 units), family and social environment (range 0-28 units), emotional state (range 0-24 units), operating capacity (range 0-28) and other concerns - bone marrow transplantation (range 0-40). The total score FACT_BMT is the sum of all the sections. Also in the subsections the higher the score the better the perceived quality of life. The physical, environmental, emotional and functional capacity is common in all FACT questionnaires used, which allows comparing this aspect between subjects.
Referred quality of life: Levels of anxiety and depression will also be assessed using the Hospital Anxiety and Depression Scale (HAD) questionnaire. (Scale info can be included in the description.) | Admission. Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  It is a self-applied questionnaire of 14 items, consisting of two subscales of 7 items, one of anxiety (odd items) and one of depression (even items). The items of the subscale of anxiety avoiding the inclusion of physical symptoms that can be confused by the patient with the symptomatology proper to his physical illness. The items on the depression subscale focus on the area of anhedonia (loss of pleasure) The score range is 0-21 for each subscale, and 0-42 for the overall score. More than 11 points for each subscale show a clinical problem. Global cutoffs are more controversial depending on the underlying disease.
Exercise tolerance | Admission. Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  measured by 6 minutes walking test
Muscle atrophy: loss or gain of weight; measured by electrical bioimpedance | Admission. Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  Gain or loss of weight with respect to the reference visit in kg.
Muscle atrophy: body mass index; measured by electrical bioimpedance | Admission. Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  Body mass index expressed in kg / m². The weight (in kg) and the height (in meters) will be used for the calculation and will be combined in the formula (weight in kg / height in m ^ 2). According to the WHO, it is considered underweight: <18.5; normal weight: 18.5-24.9; overweight: 25-29.9; degree of obesity I: 30.0-34; 5; degree of obesity II: 35.0-39.9; obesity grade III:> 40.
Muscle atrophy: fat free mass index; measured by electrical bioimpedance | Admission. Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  The fat-free mass index (kg / m²) shall be calculated as non-fat body mass (in kg) x height (in meters) ^ 2. Poor physical fitness is considered in males <18 kg / m², and in females <13.5 Kg / m².
Muscular atrophy measured by hand grip | Admission. Prior to hospital discharge or the same day discharge day. 1,3, 6, 12 months post discharge.
  Strength in the upper limbs expressed in kg.
Mortality associated to HSCT | During the HSCT process, and up to a 2-year post HSCT follow-up.
  Clinical History review.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Torralba García, RN, Principal Investigator — Hospital Clinic de Barcelona. Fundació Clinic per a la Recerca Biomédica.
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No